CLINICAL TRIAL: NCT01186159
Title: The Correlation of COX-2 Expression in Human Polymorphonuclear Leukocytes/Macrophages and Postoperative Pain
Brief Title: The Correlation of COX-2 Expression in Human Polymorphonuclear Leukocytes/Macrophages (PMNL/MP) and Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xianwei Zhang (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Xianwei Zhang, Clinical Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COX-2
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Post-Operative Pain
Keywords: COX-2; PMNL; pain; macrophages; NSAIDs
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — parecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Normal Saline (Experimental)
  Interventions: Drug: Parecoxib Sodium

INTERVENTIONS:
Drug: Parecoxib Sodium — 40 mg Parecoxib Sodium is give to the patients intravenously (diluted with 5 ml normal saline) at 30 minutes before surgery, 20 mg Parecoxib Sodium (diluted with 5 ml normal saline) at 8 hours,20 hours,32 hours,44 hours,56 hours after surgery respectively.

SUMMARY:
To investigate the dose-effect relations among the expression of COX-2 in polymorphonuclear leukocytes (PMNL) and macrophages, systemic and local inflammatory response and postoperative pain

DETAILED DESCRIPTION:
we detect COX-2mRNA, COX-2 protein expression in inflammatory cells and PGE2 concentration in patients with abdominal surgery. The differences of COX-2 expression in PMNL are compared between peripheral blood and partial incision transudate to the same individual, and at the same time, the COX-2 expression differences in PMNL and macrophages, and PGE2 concentration in partial incision transudate also compared interindividually, to show the relevance between the difference and postoperative pain. In addition, the effects of Parecoxib Sodium on COX-2 expression of the amount in PMNL and macrophages are investigated during the development of postoperative inflammatory pain. Finally, we will clear the dose-effect relations among the expression of COX-2 in inflammatory cell, systemic and local inflammatory response and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* The trial is approved by Tongji hospital's Ethics Committee, Tongji Medical College of Huazhong University of Science and Technology, and is registered through Clinical Trail. All patients give written informed consent
* American Society of Anesthesiologists (ASA) physical status of I or II
* 20 years to 55 years
* Weight 50 ~ 70 kg, BMI 19 ~ 24
* Duration of operation time in the range of 2-4 hours
* A normal leukocytes level before the operation
* No alcohol or smoking abuse
* Without major trauma, history of psychiatric disease and history of chronic pain
* Patients agreement with the trial and having ability to complete the requirements of this study
* Patients receiving intravenous patient controlled analgesia (PCA)

Exclusion Criteria:

* Allergy or contraindication to selective COX-2 inhibitors
* Received NSAIDs treatments before the operation
* Used enzyme inhibitor (such as Ketoconazole, Fluconazole, Itraconazole), enzyme inducer (such as Rifampicin, Phenytoin sodium, Carbamazepine, Dexamethasone), anticoagulant (such as Warfarin, Aspirin) and other drugs which increase the drug toxicity (such as Erythromycin, Clarithromycin, Cyclosporin Ciclosporin, ACE inhibitor or Diuretics, Lithium) from the first 3 days before the operation to postoperative observation period
* Blood transfusion, hemodilution measures in the operation
* Infection of the incision

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
COX-2 mRNA and protein expression in PMNL and macrophages without drugs intervention | 6 month
  The individual differences in COX-2 expression
the expression of COX-2 in PMNL and macrophages after the COX-2 inhibitor was used | 6 month
  The effects of COX-2 inhibitor on the expression of COX-2 in PMNL and macrophages

SECONDARY OUTCOMES:
Inflammatory mediators detection: PEG2 | 4 month
  The content of PEG2 in serum is detected by ELASA
Postoperative pain assessment | 2 month
  The visual analogue scale (VAS) at rest and patient controlled analgesia (PCA) sufentanyl consumption is assessed at all corresponding time points.

CONTACTS AND LOCATIONS:
Overall Officials: Xianwei Zhang, Doctor, Principal Investigator — Huazhong University of Science&Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China